CLINICAL TRIAL: NCT03147430
Title: Early Detection of Breast Cancer in Women With Suspicious Mammograms
Status: Active, not recruiting | Type: Observational
Sponsor: Sentara Norfolk General Hospital (Other)
Collaborators: Dorothy G. Hoefer Foundation (Other); George Mason University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-09-EX-0146
Record Dates: First submitted 2017-05-01; First posted 2017-05-10 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surgical tissue specimen slides, blood and saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Invasive Cancer: Invasive cancer confirmed by biopsy
  Interventions: Other: Biomarkers
- Benign or pre-invasive lesion: Benign or pre-invasive lesion confirmed by biopsy
  Interventions: Other: Biomarkers

INTERVENTIONS:
Other: Biomarkers — Experimentally discover putative plasma markers for detecting early, stage I breast cancer in the setting of a suspicious mammogram and distinguish those cancers from benign lesions b) verify the putative markers through molecular profiling; and c) validate the markers by mass spectrometry.

SUMMARY:
This is a non-treatment study. It will not involve the use of any investigational drug or device. Potential participants will be enrolled through direct contact with collaborating clinical sites when the patient's annual 3D mammogram report yields a BIRADS rating of 4-5. The clinical Investigators or a member of their staff will conduct consent discussion once a suspicious mammogram report is identified or if a patient is referred for imaging of a suspicious area in the breast. After consenting the participant will be asked to donate a blood sample, a saliva sample, medical records pertaining to the suspicious mammogram report and a medical history questionnaire. The participants will be followed after one year to capture progression or resolution of their suspicious mammogram report. After a biopsy confirms the diagnosis of cancer or benign lesion, a recut sample of the tissue may be requested for research.

DETAILED DESCRIPTION:
Breast cancer is a leading cause of cancer mortality in women worldwide. According to estimates, approximately 46,000 women in the United States, and 130,000 women in the European Union, die due to breast cancer yearly. Early detection is of paramount importance in reducing mortality from this major public health burden. Screening mammography has been shown to reduce breast cancer mortality by 20% to 35% in women aged 40 to 69 years. Detection of small volume breast cancer at early stages is associated with a 10-year disease-free survival rate as high as 98% in patients with pT1a,bN0M0 tumors (measuring 1 cm or less, with disease-free axillary lymph nodes and no distant metastasis). The assumption that early diagnosis will lead to improved treatment outcomes has driven the search for diagnostic biomarkers.

Despite this enthusiasm, a biomarker for stage I breast cancer has been elusive. The predictive value of mammography declines in cohorts of patients with denser breast tissue and smaller lesions, and recent studies have indicated that the small amount of biomarker molecules emanating from a breast tumor of less than 1 cm is well below the sensitivity of detection for current analytical methods. In addition, biomarkers in body fluids are highly perishable. Biomarkers break down during collection, transport and storage due to endogenous degradative enzymes yielding false negatives. Thus there is a significant need for new technologies that will a) identify and measure low abundance biomarkers (less than 1 nanogram/mL), and b) is low cost and can be seamlessly integrated into the clinical workflow.

Primary Objective:

The primary goal of this study is to a) experimentally discover putative plasma markers for detecting early, stage I breast cancer in the setting of a suspicious mammogram and distinguish those cancers from benign lesions b) verify the putative markers through molecular profiling; and c) validate the markers by mass spectrometry.

Secondary Objectives:

1. Determine percent accuracy of breast cancer diagnosis in the context of 3D mammographically (screen detected) tumors.
2. Determine percent precision of cancer diagnosis in the context of 3D mammographically (screen detected) tumors.
3. Discover additional protein markers of early stage breast cancer that distinguish these tumors from benign lesions identified by mammography by comparing protein markers between patients with invasive cancer vs. benign tumors as determined by biopsy.
4. Additionally compare protein markers between patients with invasive cancer and pre-invasive neoplasms as determined by biopsy.
5. Bank samples for future research and sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Women who receive a suspicious mammogram report or are scheduled to receive testing for suspect breast area, with a subsequent biopsy to confirm diagnosis
* Willingness and ability to donate biospecimens for the purpose of propelling research.
* Participants aged ≥ 18.

Exclusion Criteria:

* Individuals under 18 years of age or over 89 years of age.
* A known history of breast cancer.
* A diagnosis or history of any other type of cancer.
* Participants who are male.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who receive a suspicious mammogram report for breast cancer
Study Population: All participants will be enrolled through direct contact with collaborating clinical sites. In the first phase this study will strive to enroll 150 participants who are identified as having a suspicious mammogram. Review of the data for the first set of 150 patients revealed a set of biomarkers discovered and evaluated blindly that showed a strong statistical correlation with cancer versus non cancer in the final pathologic diagnosis. Based on this success, a decision is made by the PI to extend the study to enroll an additional 120 patients.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify markers to differentiate cancers from benign lesions | Duration of Study, estimated 2 years
  Experimentally discover putative plasma markers for detecting early, stage I breast cancer in the setting of a suspicious mammogram and distinguish those cancers from benign lesions, verify the putative markers through molecular profiling; and validate the markers by mass spectrometry.

SECONDARY OUTCOMES:
Determine Accuracy | 1 week (from mammogram to biospy)
  1. Determine percent accuracy of breast cancer diagnosis in the context of 3D mammographically (screen detected) tumors.
Determine Precision | 1 week (from mammogram to biospy)
  2. Determine percent precision of cancer diagnosis in the context of 3D mammographically (screen detected) tumors.
Discover additional protein markers | Duration of Study, estimated 2 years
  3. Discover additional protein markers of early stage breast cancer that distinguish these tumors from benign lesions identified by mammography by comparing protein markers between patients with invasive cancer vs. benign tumors as determined by biopsy.
Compare protein markers | Duration of Study, estimated 2 years
  4. Additionally compare protein markers between patients with invasive cancer and pre-invasive neoplasms as determined by biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hoefer, DO, Principal Investigator — Sentara Healthcare
Locations (2):
- United States (2):
  - Dorothy G Hoefer Comprehensive Breast Center, Newport News, Virginia
  - Sentara Norfolk General Breast Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No